CLINICAL TRIAL: NCT06859333
Title: An Open-label Study of the Safety, Tolerability, and Pharmacokinetic Profile of Ascending Doses of Ingavirin Forte, Capsules, Folliwing Single and Subsequent Multiple Oral Administration in Healthy Volunteers
Brief Title: Study of the Safety, Tolerability, and Pharmacokinetic Profile of Ascending Doses of Ingavirin Forte, Capsules, Folliwing Single and Subsequent Multiple Oral Administration in Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Valenta Pharm JSC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: IFR-01-01-2024
Record Dates: First submitted 2025-02-20; First posted 2025-03-05 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Influenza; Viral Respiratory Infection
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single and multiple doses, 90 mg + 5 mg (Experimental): Ingavirin Forte, 1 capsule (90 mg + 5 mg) taken once under fasted conditions, followed by Ingavirin Forte, 1 capsule (90 mg + 5 mg) taken twice a day for 2 days (the first dose under fasted conditions, the second dose under fed conditions - 2 hours after a meal), and once in the morning under fasted conditions on the 3rd day. Wash-out period after a single-dose period will last from 7 to 21 days.
  Interventions: Drug: Combined preparation of imidazolylethylamide of pentanedioic acid and N,N'-bis-[2-(1,3-diazocyclopenta-2,4-dien-4-yl)ethyl] diamide of malonic acid, 90 mg + 5 mg
- Single and multiple doses, 90 mg + 10 mg (Experimental): Ingavirin Forte, 1 capsule (90 mg + 10 mg) taken once under fasted conditions, followed by Ingavirin Forte, 1 capsule (90 mg + 10 mg) taken twice a day for 2 days (the first dose on an under fasted conditions, the second dose under fed conditions - 2 hours after a meal), and once in the morning under fasted conditions on the 3rd day. Wash-out period after a single-dose period will last from 7 to 21 days.
  Interventions: Drug: Combined preparation of imidazolylethylamide of pentanedioic acid and N,N'-bis-[2-(1,3-diazocyclopenta-2,4-dien-4-yl)ethyl] diamide of malonic acid, 90 mg + 10 mg
- Single and multiple doses, 90 mg + 20 mg (Experimental): Ingavirin Forte, 1 capsule (90 mg + 20 mg) taken once under fasted conditions, followed by Ingavirin Forte, 1 capsule (90 mg + 20 mg) taken twice a day for 2 days (the first dose under fasted conditions, the second dose under fed conditions - 2 hours after a meal), and once in the morning under fasted conditions on the 3rd day. Wash-out period after a single-dose period will last from 7 to 21 days.
  Interventions: Drug: Combined preparation of imidazolylethylamide of pentanedioic acid and N,N'-bis-[2-(1,3-diazocyclopenta-2,4-dien-4-yl)ethyl] diamide of malonic acid, 90 mg + 20 mg

INTERVENTIONS:
Drug: Combined preparation of imidazolylethylamide of pentanedioic acid and N,N'-bis-[2-(1,3-diazocyclopenta-2,4-dien-4-yl)ethyl] diamide of malonic acid, 90 mg + 5 mg — Capsules, containing 90 mg of imidazolylethylamide of pentanedioic acid and 5 mg of N,N'-bis-[2-(1,3-diazocyclopenta-2,4-dien-4-yl)ethyl] diamide of malonic acid
  Arms: Single and multiple doses, 90 mg + 5 mg
Drug: Combined preparation of imidazolylethylamide of pentanedioic acid and N,N'-bis-[2-(1,3-diazocyclopenta-2,4-dien-4-yl)ethyl] diamide of malonic acid, 90 mg + 10 mg — Capsules, containing 90 mg of imidazolylethylamide of pentanedioic acid and 10 mg of N,N'-bis-[2-(1,3-diazocyclopenta-2,4-dien-4-yl)ethyl] diamide of malonic acid
  Arms: Single and multiple doses, 90 mg + 10 mg
Drug: Combined preparation of imidazolylethylamide of pentanedioic acid and N,N'-bis-[2-(1,3-diazocyclopenta-2,4-dien-4-yl)ethyl] diamide of malonic acid, 90 mg + 20 mg — Capsules, containing 90 mg of imidazolylethylamide of pentanedioic acid and 20 mg of N,N'-bis-[2-(1,3-diazocyclopenta-2,4-dien-4-yl)ethyl] diamide of malonic acid
  Arms: Single and multiple doses, 90 mg + 20 mg

SUMMARY:
This is a Single Center, First-in-human Study of Safety, Tolerability, and Pharmacokinetic Profile of Ascending Single and Multiple Doses of Ingavirin Forte, Capsules in Healthy Volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form by the healthy subject prior to any study activities.
2. Males and females aged 18 to 45 years (inclusive) of Caucasian race.
3. Verified "healthy" diagnosis (no abnormalities detected based on clinical, laboratory, and instrumental examination methods specified in the protocol).
4. Blood pressure (BP) levels: systolic blood pressure (SBP) from 100 to 130 mm Hg (inclusive), diastolic blood pressure (DBP) from 70 to 85 mm Hg (inclusive).
5. Heart rate (HR) from 60 to 89 beats per minute (inclusive).
6. Respiratory rate (RR) from 12 to 20 breaths per minute (inclusive).
7. Body temperature from 36.0°C to 36.9°C (inclusive).
8. Body mass index (BMI): 18.5 kg/m² ≤ BMI ≤ 30 kg/m², with a minimum body weight of ≥ 55 kg for men and ≥ 45 kg for women.
9. Agreement to use adequate contraceptive methods throughout the study and for 30 days after its completion; for women of childbearing potential - a negative urine pregnancy test result.

Non-inclusion criteria:

1. Known allergic history.
2. Hypersensitivity to imidazolylethylamide of pentanedioic acid and N,N'-bis-[2-(1,3-diazocyclopent-2,4-dien-4-yl)ethyl] diamide of malonic acid (XC9) and/or excipients included in the study drug in the medical history.
3. Drug intolerance to imidazolylethylamide of pentanedioic acid and N,N'-bis-[2-(1,3-diazocyclopent-2,4-dien-4-yl)ethyl] diamide of malonic acid (XC9) and/or excipients included in the study drug.
4. Lactose intolerance, lactase deficiency, glucose-galactose malabsorption.
5. Evidence or history of chronic diseases of the kidneys, liver, gastrointestinal tract (GIT), cardiovascular, lymphatic, respiratory, nervous, endocrine, musculoskeletal, urogenital, and immune systems, as well as skin, hematopoietic and vision organs.
6. History of GIT surgery (except for appendectomy at least 1 year prior to screening).
7. Diseases/conditions that, in the judgment of the investigator, may affect the absorption, distribution, metabolism, or excretion of the study drug (SD).
8. Acute infectious diseases less than 4 weeks before screening.
9. Use of drugs that significantly affect hemodynamics, drugs affecting liver function (barbiturates, omeprazole, cimetidine, etc.), drugs that prolong the QT interval (antipsychotics (haloperidol, quetiapine, olanzapine, risperidone, sulpiride), antidepressants (fluoxetine, sertraline), antiarrhythmics (amiodarone), antibiotics (clarithromycin, azithromycin, moxifloxacin, levofloxacin, ciprofloxacin), antifungals (fluconazole), diuretics (furosemide)), less than 2 months before screening.
10. Regular use of drugs less than 2 weeks before screening and single use of drugs less than 7 days before screening (including over-the-counter drugs, vitamins, dietary supplements, herbal medicines).
11. Blood or plasma donation within 3 months before screening.
12. Use of hormonal contraceptives (in women) within 2 months before the start of screening.
13. Use of depot injections of any drugs less than 3 months before the start of screening.
14. Pregnancy or lactation; positive urine pregnancy test for women of childbearing potential.
15. Women of childbearing potential who have had unprotected sexual intercourse within 30 days prior to taking study medications with an unsterilized partner.
16. Participation in another clinical trial less than 3 months prior to screening or concurrently with this study.
17. Consumption of more than 10 units of alcohol per week in the last month before inclusion in the study or a history of alcoholism, drug addiction, or substance abuse.
18. Smoking more than 10 cigarettes per day currently or having smoked that amount in the past 6 months prior to screening; unwillingness to refrain from smoking during their stay at the research center.
19. Consumption of alcohol, caffeine, and xanthine-containing products within 7 days prior to taking the study drug.
20. Consumption of citrus fruits, cranberries, rose hips and products containing them, preparations or products containing St. John's wort within 7 days prior to taking the study drug.
21. Dehydration due to diarrhea, vomiting or other causes within the last 24 hours before taking the study drug.
22. Positive blood test to human immunodeficiency virus (HIV) types 1 and 2; antibodies to Treponema pallidum antigens; surface antigen of hepatitis B virus (HBsAg); antibodies to hepatitis C virus antigens at screening.
23. Clinically significant deviations on electrocardiogram (ECG) in medical history and/or at screening including: QTcF interval (corrected by Fredericia) ≥430 ms in men and ≥450 ms in women.
24. Information on risk factors for developing torsades de pointes such as heart failure, hypokalemia, family history of prolonged QT syndrome.
25. Positive urine test for narcotic substances and potent medications at screening.
26. Positive test for alcohol vapors at screening.
27. Planning hospitalization during the study period for any reason other than hospitalization provided for by this protocol.
28. Inability or unwillingness to comply with protocol requirements, perform procedures prescribed by the protocol, adhere to dietary and activity regimens.
29. Belonging to a vulnerable group of volunteers: students from higher and secondary medical, pharmaceutical and dental educational institutions; junior staff from clinics and laboratories; employees of pharmaceutical companies; military personnel and prisoners; individuals in nursing homes; low-income and unemployed individuals; representatives of national minorities; homeless individuals; refugees; individuals under guardianship or custody; individuals unable to give consent; as well as law enforcement officers.
30. Other conditions that, in the judgment of the investigator, may interfere with participation in the study or may lead to early withdrawal of the volunteer including adherence to fasting or special diets (e.g., vegetarianism, veganism, salt restriction) or a special lifestyle (night work hours, extreme physical exertion).

Exclusion Criteria:

1. The volunteer's withdrawal from further participation in the study.
2. Non-compliance by the volunteer with the study participation rules (missed study procedures, self-administration of prohibited medications, violation of dietary and lifestyle restrictions, etc.).
3. The emergence of reasons/situations during the study that threaten the safety of the volunteer (e.g., hypersensitivity reactions, etc.).
4. Volunteers selected for participation in the study who do not meet inclusion/exclusion criteria.
5. Development of a severe adverse event (SAE) and/or serious adverse reaction (SAR) in the volunteer during the study.
6. The volunteer requires or undergoes treatment that may affect the pharmacokinetics of the study drug.
7. Missing two or more consecutive blood samples or three or more blood samples during one study period.
8. The occurrence of vomiting/diarrhea within 8 hours after taking the study drug.
9. Positive urine test for narcotic substances and potent medications.
10. Positive test for alcohol vapors.
11. Positive pregnancy test in female participants.
12. The emergence of other reasons during the study that prevent the conduct of the study according to the protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics - Cmax | From 0 to 24 hours (single dose); from 48 to 72 hours (multiple dose)
  Maximum plasma concentration (Cmax) of imidazolylethylamide of pentanedioic acid and N,N'-bis-[2-(1,3-diazocyclopent-2,4-dien-4-yl)ethyl] diamide of malonic acid. The same analytes would be used for other pharmacokinetic measures listed below.
Pharmacokinetics - tmax | From 0 to 24 hours (single dose); from 48 to 72 hours (multiple dose)
  Time to reach Cmax (tmax)
Pharmacokinetics - AUC0-t | From 0 to 24 hours (single dose); from 48 to 72 hours (multiple dose)
  Area under the plasma concentration-time curve from time 0 to t (AUC0-t)
Pharmacokinetics - AUC0-inf | From 0 hours extrapolated to infinity after single dose and from 48 hours extrapolated to infinity after multiple dose
  Area under the plasma concentration-time curve from time 0 to infinity (AUC0-inf)
Pharmacokinetics - AUCextr | From 0 hours extrapolated to infinity after single dose and from 48 hours extrapolated to infinity after multiple dose
  Extrapolated AUC defined as (AUC0-inf - AUC0-t)/AUC0-inf
Pharmacokinetics - t1/2 | From 0 to 24 hours (single dose); from 48 to 72 hours (multiple dose)
  Elimination half-life (t1/2)
Pharmacokinetics - kel | From 0 to 24 hours (single dose); from 48 to 72 hours (multiple dose)
  Elimination constant (kel)
Pharmacokinetics - MRT | From 0 to 24 hours (single dose); from 48 to 72 hours (multiple dose)
  Mean residence time (MRT)
Pharmacokinetics - Vd | From 0 to 24 hours (single dose); from 48 to 72 hours (multiple dose)
  Volume of distribution
Pharmacokinetics - CL | From 0 to 24 hours (single dose); from 48 to 72 hours (multiple dose)
  Clearance (CL)
Pharmacokinetics - number of terminal timepoints | From 0 to 24 hours (single dose); from 48 to 72 hours (multiple dose)
  Number of points in the terminal logarithmic phase used to estimate the terminal elimination rate constant
Pharmacokinetics - AUC0-tau | From 0 to 48 hours (multiple dose)
  Steady state area under the plasma concentration-time curve from time 0 to t (AUC0-tau)
Pharmacokinetics - Cmax,ss | From 0 to 48 hours (multiple dose)
  Steady state maximum plasma concentration (Cmax,ss)
Pharmacokinetics - tmax,ss | From 0 to 48 hours (multiple dose)
  Steady state time to reach Cmax,ss (tmax,ss)
Pharmacokinetics, urine - Aeinterval | From 48 to 72 hours (multiple dose)
  The amount of active substance excreted in urine during each time interval (Aeinterval), calculated as the concentration in urine multiplied by the volume of urine.
Pharmacokinetics, urine - Ae(0-t) | From 48 to 72 hours (multiple dose)
  Total urinary excretion from zero to time t (Ae(0-t)), calculated as the sum of the amounts excreted during each time interval
Pharmacokinetics, urine - Rmax | From 48 to 72 hours (multiple dose)
  Maximum rate of urinary excretion (Rmax), calculated by dividing the amount of active substance excreted during each time interval by the time over which it was collected
Pharmacokinetics, urine - TRmax | From 48 to 72 hours (multiple dose)
  Time of maximum urinary excretion (TRmax), calculated as the average time interval during which Rmax was observed
Pharmacokinetics, urine - Fe0-t | From 48 to 72 hours (multiple dose)
  Fraction (% of dose) excreted from the body unchanged (Fe0-t), calculated as Ae/orally administered dose
Pharmacokinetics, urine - CLR | From 48 to 72 hours (multiple dose)
  Renal clearance (CLR), calculated as the ratio of Ae(0-t) to AUC(0-t)

SECONDARY OUTCOMES:
Adverse event type | From Day -14 to Day -1 (screening), from Day 1 to Day 21 (single dosing and subsequent wash-out period), from Day 1 to Day 11 (multiple dosing and subsequent observation period)
  Adverse events will be assessed by complaints, results of physical examination, results of heart rate and blood pressure assessment, results of respiratory rate assessment, body temperature, laboratory monitoring (clinical blood count, biochemical blood count, urinalysis), electrocardiography; adverse events will be classified in accordance to MedDRA.
Adverse event number | From Day -14 to Day -1 (screening), from Day 1 to Day 21 (single dosing and subsequent wash-out period), from Day 1 to Day 11 (multiple dosing and subsequent observation period)
  Number of adverse events registered during the study
Adverse event severety | From Day -14 to Day -1 (screening), from Day 1 to Day 21 (single dosing and subsequent wash-out period), from Day 1 to Day 11 (multiple dosing and subsequent observation period)
  Severity of adverse events registered during the study
Drop-outs associated with adverse events | From Day -14 to Day -1 (screening), from Day 1 to Day 21 (single dosing and subsequent wash-out period), from Day 1 to Day 11 (multiple dosing and subsequent observation period)
  The number of cases of early termination of participation in the study due to the development of adverse events and/or serious adverse events associated with the study drug
Safety and Tolerability: volunteer complaints | From Day -14 to Day -1 (screening), from Day 1 to Day 21 (single dosing and subsequent wash-out period), from Day 1 to Day 11 (multiple dosing and subsequent observation period)
  Description of any health-related complaints received from volunteer
Safety and Tolerability: physical examination results - cardiovascular system | Screening, Day 1 and 2 (single dosing), Day 1 to 4, 11 (multiple dosing)
  An assessment of the condition of the cardiovascular system and associated symptoms on physical examination (normal condition or a description of abnormal conditions/cardiovascular symptoms, if any)
Safety and Tolerability: physical examination results - respiratory system | Screening, Day 1 and 2 (single dosing), Day 1 to 4, 11 (multiple dosing)
  An assessment of the condition of the respiratory system and associated symptoms on physical examination (normal condition or a description of abnormal conditions/respiratory symptoms, if any)
Safety and Tolerability: physical examination results - digestive tract | Screening, Day 1 and 2 (single dosing), Day 1 to 4, 11 (multiple dosing)
  An assessment of the condition of the digestive tract and associated symptoms on physical examination (normal condition or a description of abnormal conditions/digestive tract symptoms, if any)
Safety and Tolerability: physical examination results - endocrine system | Screening, Day 1 and 2 (single dosing), Day 1 to 4, 11 (multiple dosing)
  An assessment of the condition of the endocrine system and associated symptoms on physical examination (normal condition or a description of abnormal conditions/endocrine symptoms, if any)
Safety and Tolerability: physical examination results - musculoskeletal system | Screening, Day 1 and 2 (single dosing), Day 1 to 4, 11 (multiple dosing)
  An assessment of the condition of the musculoskeletal system and associated symptoms on physical examination (normal condition or a description of abnormal conditions/musculoskeletal symptoms, if any)
Safety and Tolerability: physical examination results - nervous system | Screening, Day 1 and 2 (single dosing), Day 1 to 4, 11 (multiple dosing)
  An assessment of the condition of the nervous system and associated symptoms on physical examination (normal condition or a description of abnormal conditions/neurological symptoms, if any)
Safety and Tolerability: physical examination results - sensory systems | Screening, Day 1 and 2 (single dosing), Day 1 to 4, 11 (multiple dosing)
  An assessment of the condition of the sensory systems and associated symptoms on physical examination (normal condition or a description of abnormal conditions/symptoms, if any
Safety and Tolerability: physical examination results - skin/visible mucous membranes | Screening, Day 1 and 2 (single dosing), Day 1 to 4, 11 (multiple dosing)
  An assessment of the condition of the skin/visible mucous membranes and associated symptoms on physical examination (normal condition or a description of abnormal conditions/symptoms, if any)
Safety and Tolerability: vital signs - systolic blood pressure | Screening, Day 1 to 2 (single dosing), Day 1 to 4, 11 (multiple dosing)
  Systolic blood pressure (SBP, mmHg)
Safety and Tolerability: vital signs - diastolic blood pressure | Screening, Day 1 to 2 (single dosing), Day 1 to 4, 11 (multiple dosing)
  Diastolic blood pressure (DBP, mmHg)
Safety and Tolerability: vital signs - heart rate | Screening, Day 1 to 2 (single dosing), Day 1 to 4, 11 (multiple dosing)
  Heart rate (HR, bpm)
Safety and Tolerability: vital signs - body temperature (Celsius temperature scale) | Screening, Day 1 to 2 (single dosing), Day 1 to 4, 11 (multiple dosing)
  Body temperature (Celsius temperature scale)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - heart rate | Screening, Day 1 to 2 (single dosing), Day 1 to 4, 11 (multiple dosing)
  12-lead ECG (I, II, III, aVR-enhanced unipolar abduction from the right arm , aVL-enhanced unipolar abduction from the left arm, aVF - enhanced unipolar abduction from the left leg, V1-V6) taken while lying down: heart rate (beats per minute)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - PQ interval | Screening, Day 1 to 2 (single dosing), Day 1 to 4, 11 (multiple dosing)
  12-lead ECG (I, II, III, aVR-enhanced unipolar abduction from the right arm , aVL-enhanced unipolar abduction from the left arm, aVF - enhanced unipolar abduction from the left leg, V1-V6) taken while lying down: PQ interval (is the period, measured in milliseconds, that extends from the beginning of the P wave (the onset of atrial depolarization) until the beginning of the QRS complex)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - QRS complex | Screening, Day 1 to 2 (single dosing), Day 1 to 4, 11 (multiple dosing)
  12-lead ECG (I, II, III, aVR-enhanced unipolar abduction from the right arm , aVL-enhanced unipolar abduction from the left arm, aVF - enhanced unipolar abduction from the left leg, V1-V6) taken while lying down: QRS complex (the QRS complex is the combination of three of the graphical deflections seen on a typical electrocardiogram)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - corrected QT interval | Screening, Day 1 to 2 (single dosing), Day 1 to 4, 11 (multiple dosing)
  12-lead ECG (I, II, III, aVR-enhanced unipolar abduction from the right arm , aVL-enhanced unipolar abduction from the left arm, aVF - enhanced unipolar abduction from the left leg, V1-V6) taken while lying down: corrected QT interval (distance from the beginning of the QRS complex to the end of the T wave; Fredericia correction)
Safety and Tolerability: clinical blood test - hemoglobin | Screening, Day 1 and 2 (single dosing), Day 1, 3, 4, 11 (multiple dosing)
  Hemoglobin (g/L)
Safety and Tolerability: clinical blood test - hematocrit | Screening, Day 1 and 2 (single dosing), Day 1, 3, 4, 11 (multiple dosing)
  Hematocrit (%)
Safety and Tolerability: clinical blood test - red blood cell count | Screening, Day 1 and 2 (single dosing), Day 1, 3, 4, 11 (multiple dosing)
  Red blood cell count (cells/L)
Safety and Tolerability: clinical blood test - platelet count | Screening, Day 1 and 2 (single dosing), Day 1, 3, 4, 11 (multiple dosing)
  Platelet count (cells/L)
Safety and Tolerability: clinical blood test - leukocyte count | Screening, Day 1 and 2 (single dosing), Day 1, 3, 4, 11 (multiple dosing)
  Leukocyte count (cells/L)
Safety and Tolerability: clinical blood test - erythrocyte sedimentation rate | Screening, Day 1 and 2 (single dosing), Day 1, 3, 4, 11 (multiple dosing)
  Erythrocyte sedimentation rate (mm/h)
Safety and Tolerability: clinical blood test - myelocytes | Screening, Day 1 and 2 (single dosing), Day 1, 3, 4, 11 (multiple dosing)
  Leukocyte formula (myelocytes, %)
Safety and Tolerability: clinical blood test - band neutrophils | Screening, Day 1 and 2 (single dosing), Day 1, 3, 4, 11 (multiple dosing)
  Leukocyte formula (band neutrophils, %)
Safety and Tolerability: clinical blood test - segmented neutrophils | Screening, Day 1 and 2 (single dosing), Day 1, 3, 4, 11 (multiple dosing)
  Leukocyte formula (segmented neutrophils, %)
Safety and Tolerability: clinical blood test - eosinophils | Screening, Day 1 and 2 (single dosing), Day 1, 3, 4, 11 (multiple dosing)
  Leukocyte formula (eosinophils, %)
Safety and Tolerability: clinical blood test - basophils | Screening, Day 1 and 2 (single dosing), Day 1, 3, 4, 11 (multiple dosing)
  Leukocyte formula (basophils, %)
Safety and Tolerability: clinical blood test - monocytes | Screening, Day 1 and 2 (single dosing), Day 1, 3, 4, 11 (multiple dosing)
  Leukocyte formula (monocytes, %)
Safety and Tolerability: clinical blood test - lymphocytes | Screening, Day 1 and 2 (single dosing), Day 1, 3, 4, 11 (multiple dosing)
  Leukocyte formula (lymphocytes, %)
Safety and Tolerability: urinalysis - specific gravity | Screening, Day 2 (single dosing), Day 4, 11 (multiple dosing)
  Specific gravity of the urine
Safety and Tolerability: urinalysis - color | Screening, Day 2 (single dosing), Day 4, 11 (multiple dosing)
  Color of the urine
Safety and Tolerability: urinalysis - transparency | Screening, Day 2 (single dosing), Day 4, 11 (multiple dosing)
  Transparency of the urine
Safety and Tolerability: urinalysis - pH | Screening, Day 2 (single dosing), Day 4, 11 (multiple dosing)
  pH of the urine
Safety and Tolerability: urinalysis - protein | Screening, Day 2 (single dosing), Day 4, 11 (multiple dosing)
  Protein concentration (g/L)
Safety and Tolerability: urinalysis - glucose | Screening, Day 2 (single dosing), Day 4, 11 (multiple dosing)
  Glucose concentration (mmol/L)
Safety and Tolerability: urinalysis - red blood cells | Screening, Day 2 (single dosing), Day 4, 11 (multiple dosing)
  Red blood cell content (number in sight)
Safety and Tolerability: urinalysis - white blood cells | Screening, Day 2 (single dosing), Day 4, 11 (multiple dosing)
  White blood cell content (number in sight)
Safety and Tolerability: urinalysis - epithelial cells | Screening, Day 2 (single dosing), Day 4, 11 (multiple dosing)
  Epithelial cell content (number in sight)
Safety and Tolerability: urinalysis - casts | Screening, Day 2 (single dosing), Day 4, 11 (multiple dosing)
  Presence of casts (Yes/No)
Safety and Tolerability: urinalysis - mucus | Screening, Day 2 (single dosing), Day 4, 11 (multiple dosing)
  Presence of mucus (Yes/No)
Safety and Tolerability: urinalysis - bacteria | Screening, Day 2 (single dosing), Day 4, 11 (multiple dosing)
  Presence of bacteria (Yes/No)
Safety and Tolerability: urinalysis (microscopy) | Screening, Day 2 (single dosing), Day 4, 11 (multiple dosing)
  Microscopy of urine sediment is performed if it is present
Safety and Tolerability: blood chemistry - glucose | Screening, Day 1 and 2 (single dosing), Day 1 to 4, 11 (multiple dosing)
  Glucose concentration (mmol/L)
Safety and Tolerability: blood chemistry - cholesterol | Screening, Day 1 and 2 (single dosing), Day 1 to 4, 11 (multiple dosing)
  Total cholesterol concentration (mmol/L)
Safety and Tolerability: blood chemistry - protein | Screening, Day 1 and 2 (single dosing), Day 1 to 4, 11 (multiple dosing)
  Total protein concentration (g/L)
Safety and Tolerability: blood chemistry - bilirubin | Screening, Day 1 and 2 (single dosing), Day 1 to 4, 11 (multiple dosing)
  Total bilirubin concentration (micromol/L)
Safety and Tolerability: blood chemistry - creatinine | Screening, Day 1 and 2 (single dosing), Day 1 to 4, 11 (multiple dosing)
  Creatinine concentration (micromol/L)
Safety and Tolerability: blood chemistry - alkaline phosphatase | Screening, Day 1 and 2 (single dosing), Day 1 to 4, 11 (multiple dosing)
  Alkaline phosphatase activity (U/L)
Safety and Tolerability: blood chemistry - alanine transaminase | Screening, Day 1 and 2 (single dosing), Day 1 to 4, 11 (multiple dosing)
  Alanine transaminase activity (U/L)
Safety and Tolerability: blood chemistry - aspartate transaminase | Screening, Day 1 and 2 (single dosing), Day 1 to 4, 11 (multiple dosing)
  Aspartate transaminase activity (U/L)
Safety and Tolerability: blood chemistry - potassium concentration | Screening, Day 1 and 2 (single dosing), Day 1 to 4, 11 (multiple dosing)
  Potassium (mmol/L)
Safety and Tolerability: blood chemistry - sodium concentration | Screening, Day 1 and 2 (single dosing), Day 1 to 4, 11 (multiple dosing)
  Sodium concentration (mmol/L)
Safety and Tolerability: blood chemistry - chloride concentration | Screening, Day 1 and 2 (single dosing), Day 1 to 4, 11 (multiple dosing)
  Chloride concentration (mmol/L)

CONTACTS AND LOCATIONS:
Locations (1):
- State Budgetary Healthcare Institution of the City of Moscow "City Clinical Hospital No. 15 named after O.M. Filatov of the Department of Health of Moscow.", Moscow, Russia

IPD SHARING:
Plan to Share IPD: No